CLINICAL TRIAL: NCT01086696
Title: A Pilot Study of F-18 Paclitaxel (FPAC) PET for Evaluating Drug Delivery of Solid Tumors in Breast, Lung, Renal, and Adrenal Cancers
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 100078; 10-C-0078
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-05-11

CONDITIONS: Breast Cancer; Lung Cancer; Renal Cancer; Adrenal Cancer
Keywords: PET Imaging; F-18 Paclitaxel (FPAC); Breast Cancer; Lung Cancer; Renal and Adrenal Cancers; Kidney Cancer; Adrenal Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Kidney Neoplasms; Adrenal Gland Neoplasms

ARMS (2):
- 1 (Experimental): subjects with tumor types typically treatedwith taxanes
  Interventions: Drug: FPAC
- 2 (Experimental): subjects with tumor types typically treatedwith taxanes
  Interventions: Drug: FPAC

INTERVENTIONS:
Drug: FPAC — Each subject will be administered 7 mCi of FPAC,over 10-20 seconds, followed by saline flush.

SUMMARY:
Background:

* Paclitaxel is a chemotherapy drug that is commonly used to treat different types of cancers. However, cancer tumors can become resistant to paclitaxel, and as a result they will fail to accumulate sufficient concentrations of paclitaxel to kill the cancer cells. Researchers are interested in studying whether tumors have become resistant to paclitaxel, but to do so it must be possible to see how much paclitaxel is absorbed by the tumor cells.
* 18F-Fluoropaclitaxel (FPAC) is a form of paclitaxel that has been modified to be slightly radioactive in order to show up on positron emission tomography (PET) scans. By injecting a very small amount (much less that that used to treat tumors) of the radiolabeled drug into the body, researchers hope to use PET scans to evaluate the amount of the drug absorbed by solid tumors. Because FPAC is best used to study tumors located above the diaphragm, all subjects in the study will have tumors near or above the diaphragm.

Objectives:

- To determine the safety and effectiveness of FPAC as a radiological evaluation chemical.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with breast, adrenal, renal, or lung cancer and have a tumor located someone in the body at least 1 centimeter above the diaphragm.

Design:

* Participants will be screened with a physical exam, blood tests, and imaging studies as directed by the study researchers.
* Participants will receive a single dose of FPAC, followed by a series of PET scans. Regular scans will be performed for 3 hours after the dose of FPAC.
* Participants will also have a single dose of a more conventional radiotracer, followed by a series of PET scans. The results of the two sets of scans will be compared with information from previous imaging studies of participants' tumors.

DETAILED DESCRIPTION:
Background:

* Paclitaxel is a commonly used chemotherapeutic to which tumors can become resistant by failing to accumulate sufficient concentrations of the agent to be lethal to the cell.
* A noninvasive imaging test could determine the uptake of paclitaxel by tumors
* The ability to non-invasively predict chemotherapeutic uptake in solid tumors could help select patients likely to respond to treatment, estimate drug concentration within the tumor and possibly aid in the development improved of drug delivery systems and drug resistance evasion strategies.
* The PET department at the NIH developed an efficient procedure for fluorination of paclitaxel to [18F]-labeled paclitaxel (FPAC) and studied its biodistribution in rats and mice.
* Initial preclinical data shows the biodistribution of FPAC to be similar to that of paclitaxel. It is proposed that the uptake kinetics of FPAC in vivo using PET imaging will be representative of the uptake kinetics of paclitaxel
* First in human studies were performed by the PI (Kurdziel, KA) while at Virginia Commonwealth University, Richmond VA in three normal volunteers and three breast cancer patients with no adverse events. Human dosimetry estimates were obtained.
* PET/CT imaging with FPAC should permit quantitation of solid tumor uptake of the agent, which in turn should parallel paclitaxel solid tumor kinetics.
* The physiological distribution of the agent limits its use below the diaphragm. Thus, lung and breast cancers, which tend to be sensitive to taxanes, are the target tumors in this study. Adrenal and renal tumors, which tend to be insensitive to taxanes are being included as negative-control tumors.

Primary Objectives:

* Determine if the FPAC uptake in tumors is different than the uptake in normal background tissues
* Determine safety of FPAC administration

Eligibility:

* Subjects must be 18 years or older for inclusion in this study
* Subjects must have histologically proven breast, adrenal, renal or lung cancer with a lesion outside of the abdomen and pelvis greater than or equal to 1cm
* Subjects may not receive any other investigational agents 24 hours before or following FPAC injection.
* Subjects must have an ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%)
* Subjects must NOT be pregnant
* When applicable, a documented history of prior chemotherapy and radiation therapy and responses to those treatments must be available.

Design:

In this protocol, we plan to stratify enrollment into 2 groups, enrolling 15 subjects in each arm:

subjects with tumor type historically sensitive to paclitaxel therapy (lung and breast cancers) and subjects with tumor generally not responsive to paclitaxel therapy (adrenal and renal). Subjects will undergo regional dynamic FPAC PET/CT followed by static whole body imaging. All participants will undergo FDG PET/CT (outside studies permitted if submitted in DICOM format) Follow-up FDG PET/CT may be performed. (following at least 1 cycle of therapy), if applicable. If the target lesion is surgically resected, the post-treatment scan will not be performed. Subject is then expected to progress to standard or investigational therapeutic intervention (not defined by this protocol). Data regarding clinical and or imaging response to therapy will be collected if available. If a previous biopsy specimen is available, IHC for known drug transporters will also be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects must have a history of histologically or cytologically confirmed breast, lung, adrenal or renal cancer with a tumor above the diaphragm greater than or equal to 1 cm
* Subjects must be 18 years or older for inclusion in this study.
* Subjects must sign a written informed consent document and in accordance with institutional guidelines.
* If female, the subject must be postmenopausal for a minimum of two years, be surgically sterile, or have a negative pregnancy test within the 24 hours prior to tracer injection
* There are no study related limitations regarding previous radiation or chemotherapy.
* Subjects must have an ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%)
* Subjects must have normal organ and marrow function as defined below:
* leukocytes greater than or equal to 3,000/mcL
* absolute neutrophil count greater than or equal to 1,500/mcL
* platelets greater than or equal to 100,000/mcL
* total bilirubin within less than or equal to 2.5 times institutional limits OR < 3.0 mg/dl in patients with Gilbert s syndrome
* AST(SGOT)/ALT(SGPT) less than or equal to 2.5 times the institutional upper limit of normal (<5 times the ULN for patients with known hepatic metastases)
* When applicable, a documented history of prior chemotherapy and radiation therapy and responses to those treatments must be available.

EXCLUSION CRITERIA:

* Subjects may not receive any other investigational agents 24 hours prior to or following FPAC injection
* Subjects must NOT receive radiation therapy to the target lesion less than or equal to 8 weeks prior to FPAC injection
* Subjects must NOT have had surgery near the target lesion less than or equal to 4 weeks prior to FPAC injection
* Subjects with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to F-18 fluoropaclitaxel (i.e. Taxol)
* Subjects with severe claustrophobia (not relieved by oral anxiolytics) or other condition that would make them unable to lie still for the duration of the study
* Subjects with uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Subjects who are pregnant or lactating or who suspect they might be pregnant. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with FPAC, breastfeeding should be discontinued if the mother receives FPAC.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-03-09; Primary Completion 2014-08-20 (Actual); Study Completion 2016-05-11 (Actual)

PRIMARY OUTCOMES:
Uptake of FPAC in tumors | 1 hour post injection of FPAC
Safety of FPAC | 1-3 days after FPAC injection

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Kurdziel, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hsueh WA, Kesner AL, Gangloff A, Pegram MD, Beryt M, Czernin J, Phelps ME, Silverman DH. Predicting chemotherapy response to paclitaxel with 18F-Fluoropaclitaxel and PET. J Nucl Med. 2006 Dec;47(12):1995-9. PMID 17138742
- [Background] Logan J. Graphical analysis of PET data applied to reversible and irreversible tracers. Nucl Med Biol. 2000 Oct;27(7):661-70. doi: 10.1016/s0969-8051(00)00137-2. PMID 11091109
- [Background] Tang HZ. [The changes of monoamine metabolites in CSF of patients with cerebral stroke]. Zhonghua Shen Jing Jing Shen Ke Za Zhi. 1991 Jun;24(3):130-2, 186. Chinese. PMID 1716195